CLINICAL TRIAL: NCT01342250
Title: Phase Ι/Π Study of Human Umbilical Cord Mesenchymal Stem Cells Transplantation for Patients With Decompensated Liver Cirrhosis
Brief Title: Human Umbilical Cord Mesenchymal Stem Cells Transplantation for Patients With Decompensated Liver Cirrhosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen Beike Bio-Technology Co., Ltd. (Industry)
Collaborators: No.85 Hospital, Changning, Shanghai, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BKCR-LD-1.0(2010)
Record Dates: First submitted 2011-04-21; First posted 2011-04-27 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Liver Cirrhosis
Keywords: Decompensated Liver Cirrhosis; Umbilical Cord Mesenchymal Stem Cells
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Conventional plus hUC-MSCs treatment (low dose) (Experimental)
  Interventions: Biological: conventional therapy plus low dose hUC-MSCs treatment
- conventional therapy plus hUC-MSCs treatment （medium dose） (Experimental)
  Interventions: Biological: conventional therapy plus medium dose hUC-MSCs treatment
- conventional therapy plus hUC-MSCs treatment （high dose） (Experimental)
  Interventions: Biological: conventional therapy plus high dose hUC-MSCs treatment

INTERVENTIONS:
Biological: conventional therapy plus low dose hUC-MSCs treatment — patients will receive the conventional therapy plus low dose hUC-MSCs treatment
  Arms: Conventional plus hUC-MSCs treatment (low dose)
Biological: conventional therapy plus medium dose hUC-MSCs treatment — patients will receive conventional therapy plus medium dose hUC-MSCs treatment
  Arms: conventional therapy plus hUC-MSCs treatment （medium dose）
Biological: conventional therapy plus high dose hUC-MSCs treatment — patients will receive conventional therapy plus high dose hUC-MSCs treatment
  Arms: conventional therapy plus hUC-MSCs treatment （high dose）

SUMMARY:
Although liver transplantation provide a option to cure patients suffering with decompensated liver cirrhosis this condition, lack of donors, postoperative complications, especially rejection, and high cost limit its application. Bone marrow derived mesenchymal stem cells (BM-MSCs) have been shown to replace hepatocytes in injured liver, effectively rescued experimental liver failure and contributed to liver regeneration, which suggest the novel and promising therapeutic strategy In this study, the safety and efficacy of human umbilical cord mesenchymal stem cells (hUC-MSCs) transplantation for patients with decompensated liver cirrhosis will be evaluated.

DETAILED DESCRIPTION:
To investigate the safety and efficacy of human umbilical cord mesenchymal stem cells transplantation in patients of decompensated liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Aged 18-70 years.
* Decompensated liver cirrhosis, Child-Pugh B/C (7-12 points); or Meld score≦21.
* Expecting lifetime is over 2 months.
* Hepatitis B decompensated liver cirrhosis patients need antiviral therapy.

Exclusion Criteria:

* Severe drug allergic history or anaphylaxis.
* Severe problems in other vital organs(e.g. the heart, renal or lungs)
* Severe problems in psychiatric disease,such as Schizophrenia,et al
* Severe bacteria infection.
* Malignancies.
* Alcoholism or drug abuse.
* Plan to have liver transplantation in 3 months.
* Pregnancy
* Candidates who are participating in other study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | 1 year after treatment

SECONDARY OUTCOMES:
Liver function improvement | 1 year after treatment
The size of liver and the width of portal venous | 1 year after treatment
Incidence of hepatocellular carcinoma within 1 year | 1 year after treatment
Child-Pugh score, MELD score,SF36-quality of life (SF36-QOL) | 1 year after treatment
The clinical symptom improvement(including appetite, debilitation, abdominal distension, edema of lower limbs, et al ) | 1 year after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Chengwei Chen, Principal Investigator — No.85 Hospital, Changning, Shanghai, China
Locations (1):
- Shanghai Liver Disease Research Center, the Nanjing Military Command (Shanghai 85 Hospital), Shanghai, Shanghai Municipality, China